CLINICAL TRIAL: NCT04112901
Title: Activity, Mobility, Social Functioning, Mental Health and Quality of Life Outcomes in Limited Mobility Transfemoral and Knee Disarticulation Amputees Using Microprocessor-Controlled Knees or Non-Microprocessor Controlled Knees in the United Kingdom: A Cohort Study
Brief Title: Effects of Microprocessor-controlled Knee Joints on Community Outcomes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Derby (Other)
Responsible Party: Principal Investigator, Reza Safari, Research Fellow, University of Derby
Other Study IDs: V1.2
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: People With Trans-femoral Amputation
Keywords: Trans-femoral amputation; Limb prosthesis; Microprocessor Controlled Knee Joints; Community Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People with trans-femoral amputation or knee dis-articulation: include individuals with unilateral transfemoral amputation or knee disarticulation, with ≤ K2 mobility grade OR SIGAM grade D or below; i.e. able to walk ≤ 50 meters on level ground, who have been users of either microprocessor-controlled knee or non-microprocessor-controlled knee joint for at least 6 months prior to the recruitment date.
  Interventions: Device: Microprocessor-controlled knee joints; Device: Non-microprocessor-controlled knee joints

INTERVENTIONS:
Device: Microprocessor-controlled knee joints — Any type of microprocessor-controlled knee joints will be considered; this includes those controlling stance phase only (e.g. Compact C-Leg), swing phase only (e.g. Smart IP), both swing and stance phases (e.g. Reho knee), or power generating knees (e.g. POWER knee Ossur).
Device: Non-microprocessor-controlled knee joints — Any non-microprocessor-controlled knee joints such as prosthesis incorporating hydraulic, polycentric, pneumatic mechanisms, friction or locked knees.

SUMMARY:
About 21% to 35% of people with limb loss are those who lost their limb at trans-femoral level (i.e. above the knee). The increasing number of diabetes-related limb loss (amputation) and the rising proportion of older adult amputees indicates more amputees with limited mobility in the future. Among other factors, prosthesis success highly depends on the function of the knee joints during daily activities.

Presently, there are two categories of prosthetic knee joints; microprocessor-controlled knees (MPKs) and non-microprocessor-controlled knees (n-MPKs). Whilst the n-MPKs are unable to change the knee stiffness, the MPKs alter the joint stiffness and speed of movement according to the users' walking speed.

Although past studies indicate that MPKs could result in reduced risk of falls, improved balance and activity in limited mobility amputees, there is a lack of strong evidence on the effect of MPKs on community outcomes. The aim of this study is to compare activity, mobility, social functioning, depression, anxiety, and health-related quality of life in limited mobility trans-femoral or through-knee (i.e. knee disarticulation) amputees who are users of MPKs prosthesis with users of a prosthesis with n-MPKs.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transfemoral amputation or knee disarticulation
* ≤ K2 mobility grade OR SIGAM grade D or below; i.e. able to walk ≤ 50 meters on level ground,
* Users of either MPK or N-MPK for at least 6 months prior to the recruitment date.

Exclusion Criteria:

* Not meeting inclusion criteria

Ages: 18 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Amputees registered with Amputee Rehabilitation Centres across the United Kingdom.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2020-01-15 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
Short Form-36 Quality of Life (SF-36) | Baseline
  The SF-36 is a validated generic measure of health-related quality of life consisting of eight scales (physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions).

SECONDARY OUTCOMES:
Special Interest Group in Amputee Medicine (SIGAM) | Baseline
  SIGAM describe a single-item scale comprising six clinical grades (A -F) of amputee mobility. SIGAM is a self-report questionnaire with 21 dichotomous (Y/N) items and algorithm designed to facilitate grade assignment.
Prosthetic Evaluation Questionnaire (PEQ); Mobility, Social Burden and Residual Limb Health Subscales. | Baseline
  These scales contain 22 questions (Mobility and transfer, n=13; social burden, n=3, residual limb health, n=6) using the visual analog scales. The PEQ is a valid and reliable measure of the prosthetic related quality of life. It consisted of nine sub-scales, which are not dependent on each other.
Reintegration to Normal Living Index (RNLI) | Baseline
  RNLI measures the degree to which people with traumatic or incapacitating illness reintegrate into normal social activities (e.g. recreation, movement in the community, and interaction in the family or other relationships). Respondents rate 11 questions on Visual Analogue Scales.
Hospital Anxiety and Depression Scale (HADS) | Baseline
  The HADS scale is used to measure the level of anxiety and depression a person experiencing. It comprises 14 items on the four-point Likert scale; Seven items on anxiety and seven items on depression.

CONTACTS AND LOCATIONS:
Overall Officials: Reza Safari, Principal Investigator — University of Derby

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available.